CLINICAL TRIAL: NCT02350504
Title: IMPACT OF CHILDREN&Apos;S PREPARATION BEFORE MRI ON ANXIETY AND NEED FOR ANESTHESIA: A PROSPECTIVE RANDOMIZED CLINICAL TRIAL.
Brief Title: Impact of Childrens Preparation Before MRI on Anxiety and Need for Anesthesia: a Prospective Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Ilan Shelef, Department of Radiology, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SOR033614CTIL
Record Dates: First submitted 2015-01-24; First posted 2015-01-29 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Proportion of Anesthesia; Anxiety Level

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Full interactive instruction (Experimental): Full interactive instruction- which will include an instructional booklet, a movie and a simulator's practice
  Interventions: Behavioral: Full interactive instruction
- Partial instruction (Placebo Comparator): Partial instruction which included the booklet only.

INTERVENTIONS:
Behavioral: Full interactive instruction — This is a prospective randomized controlled trial in which the level of the child's exposure to instruction is controlled according to the group he is attributed to. The children are divided randomly, each Sunday (the day there is an available anesthesia staff) we change the extent of the instruction. In the intervention group, we use Full interactive instruction- which include an instructional booklet, a movie and a simulator's practice.
  Arms: Full interactive instruction

SUMMARY:
MRI has been recognized for many years as the safest and the most precise imaging method, particularly for children. However, the accuracy of MRI demands from the patient to avoid any movement while the examination is in process. This task is accomplished with difficulty by children and requires the assistance of an anesthetizing staff. In this research, our main goal is to investigate an introductory instruction as an assistive tool in performing MRI without the need in anesthesia.

DETAILED DESCRIPTION:
This is a prospective randomized controlled trial in which the level of the child's exposure to instruction is controlled according to the group he is attributed to. The children are divided randomly, each Sunday (the day there is an available anesthesia staff) we change the extent of the instruction. We use two types of instructions: 1) Full interactive instruction- which will include an instructional booklet, a movie and a simulator's practice. 2) Partial instruction which will include the booklet only.

Therefore, if it is a full instruction Sunday, all the children in that day receive full instruction and vice versa, if it will is a partial instruction Sunday, all the children in that day receive partial instruction.

All participants provide written informed consent after the study aims and procedures are fully explained.

ELIGIBILITY:
Inclusion Criteria:

* All children in the age between 5 to 16 years who come ambulatory or were hospitalized to perform an MRI test, speaks Hebrew or Arabic, are capable of understanding to their age, and their parents agreed to take part in the research

Exclusion Criteria:

* Severe cerebral palsy
* Severe ADHD
* Children that lack of communication skills

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 131 (Actual)
Dates: Start 2013-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Proportion of children which will be anesthetized | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Shelef, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

REFERENCES:
- [Background] Marshall SP, Smith MS, Weinberger E. Perceived anxiety of pediatric patients to magnetic resonance. Clin Pediatr (Phila). 1995 Jan;34(1):59-60. doi: 10.1177/000992289503400114. No abstract available. PMID 7720333
- [Background] Tyc VL, Fairclough D, Fletcher B, Leigh L, Mulhern RK. Children's distress during magnetic resonance imaging procedures. Child Health Care. 1995 Winter;24(1):5-19. doi: 10.1207/s15326888chc2401_2. PMID 10142086
- [Background] Alexander M. Managing patient stress in pediatric radiology. Radiol Technol. 2012 Jul-Aug;83(6):549-60. PMID 22763832
- [Background] de Amorim e Silva CJ, Mackenzie A, Hallowell LM, Stewart SE, Ditchfield MR. Practice MRI: reducing the need for sedation and general anaesthesia in children undergoing MRI. Australas Radiol. 2006 Aug;50(4):319-23. doi: 10.1111/j.1440-1673.2006.01590.x. PMID 16884416
- [Background] Tornqvist E, Mansson A, Hallstrom I. Children having magnetic resonance imaging: A preparatory storybook and audio/visual media are preferable to anesthesia or deep sedation. J Child Health Care. 2015 Sep;19(3):359-69. doi: 10.1177/1367493513518374. Epub 2014 Jan 31. PMID 24486815